CLINICAL TRIAL: NCT04659980
Title: Hilotherapy vs Frozen Gloves for Preventing Taxane-related Peripheral Neuropathy, Pain and Nail Toxicity in Breast Cancer
Brief Title: Preventing Taxane-related Peripheral Neuropathy, Pain and Nail Toxicity: A Prospective Self-controlled Trial Comparing Hilotherapy With Frozen Gloves in Early Breast Cancer
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universitaire Ziekenhuizen KU Leuven (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: S62794
Record Dates: First submitted 2020-12-02; First posted 2020-12-09 (Actual); Last update posted 2020-12-11 (Actual); Status verified 2020-12

CONDITIONS: Breast Cancer
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- hilotherapy (Active Comparator)
  Interventions: Device: hilotherapy
- frozen gloves (Active Comparator)
  Interventions: Device: frozen gloves

INTERVENTIONS:
Device: hilotherapy — continuous cooling of hands and feet at a constant temperature
  Arms: hilotherapy
Device: frozen gloves — cooling of hands and feet using frozen gloves
  Arms: frozen gloves

SUMMARY:
The prevention of taxane-related toxicities at the extremities is highly important for patients' treatment and quality-of-life. Unlike standard cryotherapy with frozen gloves, hilotherapy produces cooling at a constant temperature. Comparative data with frozen gloves are unavailable. This prospective self-controlled study explores the efficacy of hilotherapy at the right hand and foot compared to frozen gloves at the left in patients with early breast cancer treated with weekly paclitaxel 80 mg/m² or three-weekly docetaxel 75 mg/m².

ELIGIBILITY:
Inclusion criteria:

* adult (≥18 years) patients with breast cancer
* treated with weekly paclitaxel 80 mg/m² (12 cycles) or three-weekly docetaxel 75 mg/m² (4 or 6 cycles) in an adjuvant or neo-adjuvant setting.

Exclusion criteria:

* peripheral neuropathy or pain in the extremities at baseline, regardless of whether this was related to a prior chemotherapy treatment or another condition
* Raynaud's phenomenon, cold intolerance or any condition to the nails or peripheral blood vessels that could pose a risk to the compliance with the study interventions
* insufficient understanding of the Dutch language for self-reporting the side-effects under investigation

Patients were excluded from the analysis if they received less than two thirds of planned treatment cycles, for other reasons than the side-effects investigated in this study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 62 (Actual)
Dates: Start 2019-06-20 (Actual); Primary Completion 2020-11-20 (Actual); Study Completion 2020-11-20 (Actual)

PRIMARY OUTCOMES:
any-grade incidence of side-effects at the extremities (peripheral neuropathy, pain, nail toxicity) | 24 weeks

SECONDARY OUTCOMES:
grade 2+ side-effects at the extremities (peripheral neuropathy, pain, nail toxicities) | 24 weeks

CONTACTS AND LOCATIONS:
Locations (1):
- University Hospitals Leuven, Leuven, Belgium

IPD SHARING:
Plan to Share IPD: Undecided